CLINICAL TRIAL: NCT06420739
Title: Improving Patient Safety for Surgical Patients on Semaglutide: A Gastric Ultrasound Initiative
Brief Title: The Semaglutide Study
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5873
Record Dates: First submitted 2024-04-10; First posted 2024-05-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Fasting
Keywords: Gastric Ultrasound; Fasting; Semaglutide; Elective surgery
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gastric Ultrasound — Bedside Gastric Ultrasound to determine the volume and nature of gastric content in patients before their surgery.

SUMMARY:
The primary goal of this study is to evaluate the incidence of "full stomach" in fasting elective surgical patients on Semaglutide medication. The other goals are to study the impact of the time interval since the last dose of the medication on the incidence of full stomach and to develop evidence-based recommendations for the perioperative management of these patients.

DETAILED DESCRIPTION:
Pulmonary aspiration of gastric contents has long been recognized as a threat to anesthesia patient safety. Most elective surgical patients, however, are considered to be at low risk for this complication provided they abstain from eating solid food for at least 8 hours prior to anesthesia and for clear fluids for at least 2 hours. The recent introduction of GLP-1 agonists (such as Semaglutide), a new class of drugs for the treatment of diabetes and weight loss, has challenged the status quo, and is posing a new threat to perioperative patient safety.There are recent reports of aspiration of large amounts of particulate undigested food in the perioperative period on patients taking Semaglutide despite prolonged fasting of over 12 hours, one of those cases happening at the UHN.This is of great concern given the explosive increase in use of these medications globally.In the month of June 2023, three North American anesthesiology societies (the Canadian Anesthesiologists' Society, the American Society of Anesthesiologists and the Anesthesia Patient Safety Foundation) have raised the alert regarding an increased risk of aspiration under anesthesia while on these drugs.Given the long half-life of up to 7 days, a true reduction of risk would necessitate holding these drugs preoperatively for longer periods than are usually feasible.

Management strategies recommended to date include treating every patient on Semaglutide as if they have a 'full stomach", avoiding general anesthesia if possible and even considering surgical cancellation if the patient presents symptoms such as nausea and vomiting, which are common while on these medications. While these recommendations stand to reason, they are over-arching, targeted to all patients and could result in unnecessary surgical cancellations or invasive procedures (such as nasogastric tube insertion, endotracheal intubation and rapid sequence induction) which have their own set of risks.

This timely study addresses the current knowledge gap and a recently identified threat to perioperative patient safety that has been highlighted by three major anesthesiology societies in the past 2-3 months. Our team at the UHN is uniquely positioned to shed some light into these pressing questions and develop management recommendations that optimize safety while avoiding unnecessary surgical cancellations and targeting invasive procedures for airway management only to those patients that really need them.

Our group has previously developed and validated a simple, non-invasive bedside ultrasound test that can differentiate a safe "empty stomach" from a "full stomach" that may pose an increased risk of aspiration under anesthesia. The investigators have validated this bedside test in the adult, pediatric, obstetric and morbidly obese populations.

Hypothesis:

Patients on Semaglutide will have an increased incidence of full stomach to at least 10%, compared to a baseline of 5%, a difference that the investigators consider clinically significant.

Study design:

This is a prospective cohort study.

Study population:

The investigators propose to study a cohort of 100 patients undergoing elective surgery while under treatment with Semaglutide for either diabetes or for losing weight.

Patients who are on Semaglutide for at least a month will be identified, screened for eligibility, and invited to participate in this study.All identified patients will be given standard pre-operative fasting instructions as per current institutional practice for elective surgical patients (a minimum of 8 hours of fasting for solid food and 4 hours for clear fluids).

A bedside gastric ultrasound examination will be performed using a portable ultrasound unit and a curvilinear low-frequency probe with abdominal settings. The exam will be done in two positions (supine and right lateral decubitus). The gastric antrum will be identified in a sagittal plane in the epigastric area between the left lobe of the liver anteriorly and the pancreas and aorta posteriorly. The type of gastric content (nothing, clear fluid or solid) will be documented based on qualitative findings.

If clear fluid is present our mathematical model will be used to estimate the volume based on a cross-sectional area of the gastric antrum:

(Volume (ml) = 27.0 + 14.6 x CSA (cm2) - 1.28x age (year).11

A stomach will be considered:

1. "empty" and consistent with "low aspiration risk" if the antrum appears completely empty in both supine and right lateral decubitus position (Grade 0 antrum) or there is clear fluid with a volume < 1.5 mL/Kg which is consistent with a low-risk situation.
2. "full" or at risk of aspiration if there is any amount of solid content or clear fluid with a volume, > 1.5 mL/Kg.

The result of the gastric ultrasound study will be shared with the attending anaesthesiologist in charge of every patient who will be free to establish what they consider the safest management plan based on their clinical judgement and the ultrasound results. The surgical timing (on time, delayed or cancelled), the type of anaesthetic used, and the airway management strategies will be documented. Changes in anaesthetic management from the a priori plan will be documented. Any episodes of regurgitation or aspiration in the perioperative period will be documented. Information on anaesthetic technique, airway management and the incidence of regurgitation and aspiration throughout the intraoperative period will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective surgery at Toronto Western Hospital
2. Aged ≥ 18 years of age
3. American Society of Anaesthesia physical status classification I to III
4. Patients being treated with Semaglutide for at least 1 month

Exclusion Criteria:

1. Current pregnancy evidenced by positive urinary pregnancy test
2. Previous surgery of the upper gastrointestinal tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 100 patients undergoing elective surgery while under treatment with Semaglutide for either diabetes or for losing weight.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of full stomach. | Pre-Surgical fasting duration per guideline
  Frequency of full stomach in patients taking semaglutide and fasting before surgery. Analysis of the primary outcome will be based on a chi-square analysis.

SECONDARY OUTCOMES:
Any changes in anesthetic management from the a priori plan following the result of the gastric ultrasound examination. | Pre-operative anesthesia management plan
  The investigators will measure the frequency of changes in management plan
Impact of age, sex and the time since the last dose of Semaglutide, on the incidence of "full stomach". | Pre-Surgical fasting duration per guideline
  The investigators will compare the absolute incidence of "full stomach" in patients receiving the last dose less than 7 days before surgery with those with last dose between 7-14 days and > 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, Principal Investigator — Investigator-Sponsor
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No